CLINICAL TRIAL: NCT02666651
Title: Regional Tolvaptan Registry
Acronym: Tolvaptan
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiology Research UBC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H15-00115
Record Dates: First submitted 2016-01-14; First posted 2016-01-28 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Decompensated Heart Failure; Hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group (Experimental): Administration of oral tolvaptan (15-60mg PO titration) during admission for decompensated heart failure
  Interventions: Drug: Tolvaptan
- Control group (Other): There is no intervention planned for the Control group. Aggregate administrative regional data describing patient outcomes from the local health authority
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan is dispensed during hospitalization according to its product monograph and clinician discretion. It will be discontinued once serum sodium is normalized, or in the case of a drug related adverse event or hospital discharge.
  Other Names: Samsca
  Arms: Test group
Other: No intervention — There is no intervention planned for the Control group. Aggregate administrative regional data describing patient outcomes from the local health authority will be used as a comparator.
  Arms: Control group

SUMMARY:
Low blood sodium is a common observation in patients presenting with heart failure and is associated with increased mortality, prolonged hospital stay, and repeat hospital visits. Tolvaptan is a new and approved medication to treat low sodium levels in patients who present with symptoms of heart failure, however, it is not currently available as a treatment option due to high costs not covered by our provincial plan. In this observational, non-randomized study the drug will be provided to all subjects free of charge and given only during their hospital stay. After discharge subjects will be followed for 6 months (3 visits).

DETAILED DESCRIPTION:
Purpose: A prospective, open-label, real life registry of Tolvaptan in hospitalized heart failure patients with hyponatremia.

Hypothesis: Administration of Tolvaptan in hospitalized patients with heart failure and hyponatremia will demonstrate improvements in patient symptom status and cost savings from decreased healthcare utilization.

Justification: In clinical trials, Tolvaptan has been shown to quickly, effectively, and safely improve sodium levels in heart failure patients, and decrease the length of hospital stay and improve symptom status compared to placebo. Although Tolvaptan is an approved drug in Canada for the treatment of patients hospitalized with heart failure and hyponatremia, its availability is limited to private buyers and not available on hospital formularies due to cost constraints. There are no alternatives to this first in class agent.

Objectives: The primary endpoint is reduction in length of stay for heart failure in registry participants compared to length of stay in the Vancouver Coastal Health (VCH) administrative data set. Secondary endpoints will include recurrent hospitalization, change in quality of life, and B-type Natriuretic Peptide (BNP) levels over the study period.

Research Method: Patients admitted to Vancouver General Hospital (VGH) with heart failure and hyponatremia will be identified through clinical referral by cardiologists who have ensured that all other measures have been undertaken to improve the patient's clinical status.

Tolvaptan is dispensed according to product monograph and clinician discretion, and will be discontinued once serum sodium is normalized, or in the case of a drug related adverse event or hospital discharge. Bloodwork will be drawn to monitor liver function and electrolytes during hospitalization and in follow up. Data will be captured from time of consent until 6 months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has clinical evidence of heart failure AND elevated BNP or evidence of left ventricular dysfunction (left ventricular ejection fraction (LVEF) < 40%) on diagnostic imaging.
2. Serum sodium < 130 mmol/L OR serum sodium 131-134 mmol/L and symptomatic.
3. Sodium and fluid restriction ongoing.
4. Trial of optimal diuretic therapy (at prescribing physician's clinical discretion).
5. Discontinuation of non-essential medications/treatments that are known to cause hyponatremia.

Exclusion Criteria:

1. Life expectancy < 6 months
2. Documented adverse events with tolvaptan in the past
3. Meet exclusion criteria from the Study of Ascending Levels of Tolvaptan in Hyponatremia (SALT Trial):

   * Serum sodium < 120mmol/L if neurologic impairment
   * Confounding disease (e.g. recent stroke or myocardial infarction (MI), recent surgery, uncontrolled diabetes, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | Subjects are followed for 6 months after discharge
  Hospital length of stay for heart failure in the treatment group will be measured as days and compared to administrative regional data describing patient outcomes from the local health authority.

SECONDARY OUTCOMES:
Recurrent hospitalization. | Subjects are followed for 6 months after discharge
  This will be measured by the number of times a patient is readmitted to hospital following their discharge from the initial hospitalization.
Change in quality of life. | Subjects are followed for 6 months after discharge
  This will be assessed by administrating the Minnesota Living with Heart Failure questionnaire at initial hospitalization, 1 month follow-up, 3 month follow-up, and 6 month follow-up timepoints.
BNP (Brain-Type Natriuretic Peptide) levels | Subjects are followed for 6 months after discharge
  BNP is an established biomarker of CHF severity and blood samples will be collected at 1, 3, and 6 month visits. Values will be collected as a continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Virani, MD, MSc, MPH, FRCPC, Principal Investigator — Director of the Heart Failure and Cardiology-Oncology Programs at VGH
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided